CLINICAL TRIAL: NCT02472353
Title: A Phase II Pilot Study Using Metformin to Reduce Cardiac Toxicity in Breast Cancer Patients
Brief Title: Use of Metformin to Reduce Cardiac Toxicity in Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: did not meet target accrual
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMEM-2014-MET001
Record Dates: First submitted 2015-06-09; First posted 2015-06-15 (Estimated); Results first posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Breast Tumors
Keywords: breast; cancer; doxorubicin; metformin; cardiotoxicity; ejection fraction; LVEF
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Cardiotoxicity | interventions — Metformin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): Patients will receive standard of care for their breast cancer with no metformin during their treatment with doxorubicin.
  Interventions: Drug: Doxorubicin
- Metformin + Standard of Care (Experimental): Patients will receive metformin during their treatment with doxorubicin for their breast cancer.
  Interventions: Drug: Metformin; Drug: Doxorubicin

INTERVENTIONS:
Drug: Metformin — Metformin will begin to be administered prior to treatment with doxorubicin. Metformin will continue to be given throughout doxorubicin cycles until the completion of doxorubicin therapy.
  Other Names: Glucophage
  Arms: Metformin + Standard of Care
Drug: Doxorubicin — Standard of care treatment with doxorubicin

SUMMARY:
The goal of this study is to determine if co-administration of metformin and doxorubicin in breast cancer patients receiving neoadjuvant or adjuvant therapy will reduce the number of patients who develop a significant change in left ventricle ejection fraction (LVEF).

DETAILED DESCRIPTION:
This is a randomized, open-label, phase II design pilot study in patients with breast cancer requiring neoadjuvant or adjuvant chemotherapy. Eligible patients will be equally randomized to either receive metformin plus standard of care therapy or standard of care therapy alone. Patients receiving metformin will continue drug until the doxorubicin-containing cycles are complete, unless unacceptable toxicity occurs or the patient decides to withdraw from the study. Both arms of the study will undergo echocardiograms with contrast at baseline, upon completion of doxorubicin-containing cycles (within 28 days of completion), and at the one-year and seven-year time points. Additionally biomarker labs will be obtained to explore if there is a correlation between change in cardiac activity and the activity of metformin. If willing, all enrolled patients will provide a sample of whole blood for further exploratory analysis. Symptoms reported during the study will be correlated with know single nucleotide polymorphisms (SNPs) found during an exploratory genomic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer requiring neoadjuvant or adjuvant therapy with doxorubicin
* Complete metabolic panel demonstrating adequate organ functions as defined by the following: Aspartate transaminase (AST) less than 2.5 times Upper Limit of Normal (ULN); Alanine transaminase (ALT) less than 2.5 times ULN; alkaline phosphatase less than 2.5 times ULN; serum creatinine less than 1.5 mg/dL; serum bilirubin less than ULN
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Age greater than or equal to 21 years

Exclusion Criteria:

* Known diabetes
* History of cardiac arrhythmias or symptomatic cardiac disease
* Currently taking antiarrhythmic medications, beta-blockers, or other rate controlling cardiac medications
* Currently taking metformin and/or sulfonylureas
* Known hypersensitivity or intolerance to metformin
* Baseline ejection fraction of less than 50% measured by echocardiogram
* Known hypersensitivity to contrast used during echocardiogram
* Risk factors associated with increased risk of metformin-associated lactic acidosis (e.g. congestive heard failure, history of acidosis, habitual intake of 3 or more alcoholic beverages per day)
* Pregnant or breast feeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Williams, CNP, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Cancer Institute, Sioux Falls, South Dakota, United States

REFERENCES:
- [Derived] Sun ML, Dong JM, Liu C, Li P, Zhang C, Zhen J, Chen W. Metformin-mediated protection against doxorubicin-induced cardiotoxicity. Biomed Pharmacother. 2024 Nov;180:117535. doi: 10.1016/j.biopha.2024.117535. Epub 2024 Oct 15. PMID 39405911

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Referrals and investigator's own patients
Period: Overall Study
Arm/Group | Standard of Care | Metformin + Standard of Care
Started | 14 | 16
Completed | 10 | 10
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Study Termination | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Metformin + Standard of Care | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 0 | 4 | 4
Age, Continuous [Mean (Full Range); unit: years] | 43 [31 to 64] | 53 [29 to 68] | 53 [29 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 16 | 30
Echocardiography [Number; unit: participants] | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Less Than or Equal to 5% Decrease in Left Ventricle Ejection Fraction (LVEF) on Echocardiogram
Description: Determine whether the addition of metformin to standard doxorubicin therapy in breast cancer patients will decrease the incidence of change in left ventricle ejection fraction (LVEF).
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Metformin + Standard of Care
Number analyzed (Participants) | 10 | 10
Participants | 4 | 5

ADVERSE EVENTS:
Time Frame: Time point 1: Within 2 weeks of starting metformin Time point 2: 4 weeks after starting metformin Time point 3: 7 weeks after starting metformin Time point 4: 9 weeks after starting metformin (last assessment during treatment period)
Arm/Group | Standard of Care | Metformin + Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 3/16
Other Adverse Events (participants affected / at risk) | 12/14 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=14) | Metformin + Standard of Care (N=16)
Pain (General disorders) | 0 (0) | 1 (1) — admitted for pain control for herpes zoster outbreak
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Infection (Infections and infestations) | 0 (0) | 1 (1) — admitted for central line infection
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=14) | Metformin + Standard of Care (N=16)
Anemia (Blood and lymphatic system disorders) | 10 (17) | 14 (39)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (10) | 7 (15)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (11)
Depression (Psychiatric disorders) | 3 (4) | 3 (4)
Water Eyes (Eye disorders) | 1 (1) | 2 (2)
Hot Flashes (Vascular disorders) | 7 (8) | 10 (28)
Diarrhea (Gastrointestinal disorders) | 8 (12) | 13 (26)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Decreased Platelets (Investigations) | 2 (2) | 2 (2)
Decreased WBC (Investigations) | 4 (4) | 6 (9)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 11 (22)
Weight Loss (Investigations) | 2 (2) | 4 (6)
Tachycardia (Cardiac disorders) | 1 (1) | 4 (6)
Constipation (Gastrointestinal disorders) | 7 (12) | 7 (13)
Anxiety (Psychiatric disorders) | 6 (6) | 9 (15)
Headache (Nervous system disorders) | 6 (10) | 9 (19)
Pain (General disorders) | 9 (15) | 6 (7)
Fatigue (General disorders) | 12 (20) | 16 (49)
Insomnia (Psychiatric disorders) | 9 (12) | 10 (28)
Dysphagia (Nervous system disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
Increased AST (Investigations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Neuropathy (Nervous system disorders) | 7 (9) | 4 (7)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 5 (8)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Hypertension (Vascular disorders) | 8 (14) | 9 (12)
Nausea (Gastrointestinal disorders) | 9 (16) | 12 (29)
Oral Mucositis (Gastrointestinal disorders) | 7 (7) | 7 (10)
Fever (General disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 7 (12)
Increased ALT (Investigations) | 4 (4) | 3 (3)
Dysgeusia (Nervous system disorders) | 9 (11) | 7 (12)
Vomiting (Gastrointestinal disorders) | 3 (4) | 5 (6)
Edema (General disorders) | 1 (1) | 5 (7)
Dyspnea (Gastrointestinal disorders) | 5 (6) | 2 (6)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (8)

LIMITATIONS AND CAVEATS:
The study was terminated early due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT02472353/Prot_SAP_000.pdf